CLINICAL TRIAL: NCT05148598
Title: Scleroderma Treatment With Celution Processed Adipose Derived Regenerative Cells - A Randomized, Double-Blind, Placebo-Controlled Study - The STAR-II Trial
Brief Title: ADRCs in The Treatment of Hand Dysfunction Due to Scleroderma
Acronym: STAR-II
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Paracrine, INC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STAR-II, 2021-03.V1
Record Dates: First submitted 2021-11-20; First posted 2021-12-08 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2021-12

CONDITIONS: Scleroderma, Diffuse
Keywords: Hand Dysfunction; Scleroderma; Scleroderma, Diffuse
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: * Prospective
  * Randomized Parallel Group
  * Placebo-Controlled
  * Safety and Efficacy Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo is visually indistinguishable from active treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ADRC Arm (Experimental): Subjects in the ADRC arm will receive standard care and active treatment (ADRCs)
  Interventions: Device: ADRCs; Other: Standard Care
- Standard Care Arm (Placebo Comparator): Subjects in the Standard Care arm will receive standard care and Placebo
  Interventions: Other: Standard Care; Other: Placebo

INTERVENTIONS:
Device: ADRCs — Adipose Derived Regenerative Cells (ADRCs) processed with Celution System
  Arms: ADRC Arm
Other: Standard Care — Standard care
Other: Placebo — Placebo visually indistinguishable from ADRCs
  Arms: Standard Care Arm

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of the Celution Device in the processing of an autologous graft consisting of adipose derived regenerative cells (ADRCs) in the treatment of hand dysfunction due to scleroderma.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and efficacy of the Celution Device in the processing of an autologous graft consisting of adipose derived regenerative cells (ADRCs) in the treatment of hand dysfunction due to scleroderma.

ELIGIBILITY:
Key Inclusion Criteria:

* Diffuse cutaneous scleroderma (duration > 5 years)
* Cochin Hand Function Scale ≥ 20 units
* Symptoms consistent with Raynaud's Phenomenon
* Ability to safely undergo liposuction

Key Exclusion Criteria:

* Active infection
* Contracture(s) of any finger
* Sympathectomy within 6 months of Screening Visit
* Rheumatoid Arthritis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Cochin Hand Function Score | 26 weeks
  Cochin Hand Function Score

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available.